CLINICAL TRIAL: NCT03583151
Title: Injection With Amniotic Fluid Versus Corticosteroid in Patients With Stenosing Tenosynovitis: a Randomized, Blinded Trial
Brief Title: Corticosteroid vs. Amniotic Fluid Injections in Patients With Trigger Finger
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: J&M Shuler (Industry)
Collaborators: Vivex Biomedical (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Random TF
Record Dates: First submitted 2018-06-28; First posted 2018-07-11 (Actual); Last update posted 2018-07-11 (Actual); Status verified 2018-06

CONDITIONS: Stenosing Tenosynovitis
Keywords: Corticosteroid
MeSH Terms: conditions — Tendon Entrapment | interventions — Steroids

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Steroid injection (Active Comparator): 1 mL Solu-medrol mixed with 0.5mL marcaine and 0.5 mL of lidocaine
  Interventions: Biological: Steroid injection
- Amniotic fluid injection (Experimental): 1 mL amniotic fluid mixed with 0.5mL marcaine and 0.5 mL of lidocaine
  Interventions: Biological: Amniotic fluid injection

INTERVENTIONS:
Biological: Amniotic fluid injection — Amniotic fluid contains various proteins that support cell proliferation, movement and differentiation. Amniotic fluid also includes collagen substrates, growth factors, amino acids, polyamines, lipids, carbohydrates, cytokines, extracellular matrix molecules like hyaluronic acid and fibronectin, cells and other chemical compounds that are needed for tissue protection and repair.
  Arms: Amniotic fluid injection
Biological: Steroid injection — Solu-medrol
  Arms: Steroid injection

SUMMARY:
The proposed study aims to investigate whether amniotic fluid injections are a better alternative to corticosteroid injections as a conservative treatment for stenosing tenosynovitis. Based on results from our most recent pilot study exploring patient outcomes after receiving an amnion injection, we were able to observe symptom resolution in more than half of the study population. Adverse events were extremely rare and not related to study participation. Given the numerous occurrences of successful symptom resolution, the next step is to compare patient outcomes to those of patients who receive the standard steroid injection. This study will compare outcome measurements of patients who receive amnion injections to those who receive steroid injections.

ELIGIBILITY:
Inclusion Criteria:

* Patient is at least 18 years of age
* Patient is diagnosed with stenosing tenosynovitis

Exclusion Criteria:

* Patient is less than 18 years of age
* Pregnancy
* Enrolling clinician does not believe that the patient is mentally capable of understanding the research nature of the procedure due to mental handicap/disability or illiteracy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2018-05-10 (Actual); Primary Completion 2018-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Patient reported pain level | 12 months
  Analog pain scale (0-10)

SECONDARY OUTCOMES:
Trigger frequency | 12 months
  Rate at which a patient's digit will lock or trigger
Disabilities of the Arm Shoulder and Hand score | 12 months
  Measure of disability in performing every day activities at work and around the house. Calculated value from DASH questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Shuler, MD, Principal Investigator — Athens Orthopedic Clinic
Locations (1):
- Athens Orthopedic Clinic, Athens, Georgia, United States

IPD SHARING:
Plan to Share IPD: Undecided